CLINICAL TRIAL: NCT03151304
Title: A Two-Stage, Open-Label Phase 2 Study of Pracinostat and Azacitidine in Patients With IPSS-R High and Very High Risk Myelodysplastic Syndromes Previously Untreated With Hypomethylating Agents
Brief Title: A Safety and Efficacy Study of Pracinostat and Azacitidine in Patients With High Risk Myelodysplastic Syndromes
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor's decision as at the completion of the primary analysis, the data were considered mature
Sponsor: Helsinn Healthcare SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEI-011
Record Dates: First submitted 2017-05-05; First posted 2017-05-12 (Actual); Results first posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Myelodysplastic Syndromes
Keywords: MDS
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — SB939 compound; Azacitidine

STUDY DESIGN:
Intervention Model Description: Two-Stage, Open-Label
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Stage 1a and 1b open-label pracinostat plus azacitidine (Experimental): open-label single arm pracinostat plus azacitidine. Pracinostat: 45 mg administered orally 3 days each week for 3 consecutive weeks, followed by 1 week of rest, in 28-day cycles.
  In later cycles (i.e., after Cycle 4), pracinostat dose reduction to 45 mg orally 3 days each week × 2 weeks (instead of 3 weeks) or dose interruption is allowed to manage toxicity such as fatigue, gastrointestinal toxicity, or myelosuppression.
  Azacitidine: 75 mg/m2 for 7 days of each 28-day cycle. Administration will occur by subcutaneous (SC) injection, or IV infusion if SC injections are not tolerated, on one of two schedules:
  * Schedule 1 - daily therapy on Days 1 through 7
  * Schedule 2 - 5-2-2 schedule in which subjects receive azacitidine for 5 consecutive days (Days 1 through 5) with rest on Days 6 and 7, and resume azacitidine dosing the first two days of the next week (Days 8 and 9) of each 28-day cycle
  Interventions: Drug: Pracinostat; Drug: Azacitidine

INTERVENTIONS:
Drug: Pracinostat — 45 mg capsule
  Other Names: SB939
Drug: Azacitidine — SC or IV injection

SUMMARY:
This is a Phase 2, two-stage study of the safety and efficacy of pracinostat in combination with azacitidine in patients with IPSS-R high and very high risk myelodysplastic syndrome (MDS) who are previously untreated with hypomethylating agents (HMAs). Enrollment in this study will be limited to high/very high risk MDS because this group represents the highest unmet need, with median survival of less than 18 months.

Stage 1a will be conducted as an open-label single arm in up to 40 subjects to assess if this regimen with a lower pracinostat dose results in a discontinuation rate that meets a predefined threshold and in efficacy that justifies expansion of enrollment into Stage 1b.

A discontinuation rate of approximately ≤10% in Stage 1a, a rate comparable to that observed with azacitidine alone in study MEI-003 (NCT01873703), supports expansion into Stage 1b.

Stage 1b will be conducted as expansion of stage 1a. Approximately 20 additional subjects will be enrolled. Study drugs should be continued until disease progression or intolerable toxicity. It is important to note that the median time to achieving a response with azacitidine alone is 4 to 5 months. Furthermore, the median time to achieving a Complete Response (CR) in study MEI-003 (NCT01873703) was 4 cycles. Therefore, early (<6 months) discontinuation of trial therapy for 'no response' should be avoided. The Medical Monitor should be contacted prior to discontinuing a subject from the study to discuss the rationale for discontinuation.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male subjects ≥18 years-of-age.
2. Histologically or cytologically documented diagnosis of MDS according to the World Health Organization (WHO) classification (Vardiman 2009, Arber 2016) with >5% and <20% bone marrow blasts by morphology and a peripheral white blood cell (WBC) count of <20,000/μL

   * If WBC ≥20,000/μL, cytoreduction with hydroxyurea is permitted prior to enrollment.
   * chronic myelomonocytic leukemia CMML-1 and CMML-2 subtypes
3. Classified as high or very high risk according to the Revised International Prognostic Scoring System (IPSS-R) risk category. CMML-1 and CMML-2 subtypes will be considered high-risk MDS and will not require IPSS-r scoring
4. Bone marrow biopsy (BMBx) and/or aspirate within 28 days prior to first study treatment.
5. Clinical indication for treatment with azacitidine.
6. Previously untreated with HMAs (prior therapy with transfusions, hematopoietic growth factors, or immunosuppressive therapy is allowed).

   a. subjects who require the start of an HMA (e.g., azacitidine) due to progressing MDS may receive up to 1 cycle of azacitidine within 30 days prior to planned first dose (Cycle 1 Day 1)
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
8. Adequate organ function as evidenced by:

   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 × the upper limit of normal (ULN).
   * Total bilirubin ≤1.5 × ULN or total bilirubin of ≤2 mg/dL, whichever is higher. Total bilirubin < 3 x ULN for patients with Gilbert-Meulengracht Syndrome
   * Serum creatinine <1.5 mg/dL, or creatinine clearance>40 mL/min.
   * QTcF interval ≤450 msec using the mean of triplicate electrocardiograms (ECGs).
9. Female subjects of childbearing potential and male subjects with female partners of childbearing potential are required to use two forms of acceptable contraception, including one barrier method, during their participation in the study and for 30 days following last dose. Female subjects of childbearing potential must not be breastfeeding, or planning to breastfeed, and must have a negative pregnancy test ≤7 days before first study drug administration.

   Male subjects must also refrain from donating sperm during their participation in the study.
10. Voluntary written informed consent before performance of any study-related procedure not part of normal medical care.
11. Have the willingness and ability to understand the nature of this study and to comply with the study and follow-up procedures.

Exclusion Criteria:

1. Bone marrow blasts ≥20%, indicating a diagnosis of acute myeloid leukemia (AML).
2. Received any of the following within the specified time frame prior to administration of study medication:

   * Any investigational agent within 14 days or 5 half-lives prior to enrollment, whichever is longer.
   * Hydroxyurea within 48 hours prior to first day of study treatment.
   * Hematopoietic growth factors: erythropoietin, granulocyte colony stimulating factor (G-CSF), granulocyte macrophage colony stimulating factor (GM-CSF), or thrombopoietin receptor agonists at least 7 days (14 days for Aranesp), prior to study enrollment.
   * Major surgery within 28 days prior to first study treatment.
3. Subjects who have not recovered from side effects of previous therapy.
4. Cardiopulmonary function criteria:

   * Current unstable arrhythmia requiring treatment.
   * History of symptomatic congestive heart failure (New York Heart Association [NYHA] Class III or IV).
   * History of myocardial infarction, pulmonary embolism or cerebrovascular accident within 6 months of enrollment.
   * Current unstable angina.
5. Prior treatment for MDS with histone deacetylase (HDAC) inhibitors Zolinza (vorinostat), Belenodaq (belinostat), Farydak (panobinostat), Istodax (romidepsin/depsipetide), or investigational agent with significant action as an HDAC inhibitor.
6. Clinical evidence of central nervous system involvement.
7. Subjects with gastrointestinal (GI) tract disease causing the inability to take oral medication, malabsorption syndrome, a requirement for intravenous (IV) alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's disease, ulcerative colitis).
8. Uncontrolled infection with human immunodeficiency virus (HIV) or chronic hepatitis B or C.
9. Life-threatening illness unrelated to cancer or any serious medical or psychiatric illness that could, in the Investigator's opinion, potentially interfere with participation in this study.
10. Presence of a malignant disease within the last 12 months, with the exception of adequately treated in-situ carcinomas, basal or squamous cell carcinoma, non-melanomatous skin cancer, or malignancies treated with curative intent and no evidence of active disease in prior 12 months and felt to be low risk for recurrence. Other malignancies may be considered after consultation with the Medical Monitor
11. An unwillingness or inability (including breastfeeding women, prohibited concomitant medications, uncontrolled infections, psychological, familial, sociological, or geographical conditions) to comply with study and/or follow-up procedures as outlined in the protocol
12. Known hypersensitivity to any components of pracinostat, azacitidine or mannitol
13. Current smoking or vaporizing of tobacco or cannabis-related products (use of patches, chewing tobacco, or nicotine gum is permitted). Subjects who stopped smoking at least 8 days prior to first pracinostat dosing can be, provided they refrain from smoking during the whole study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Ghalie, MD, Study Director — MEI Pharma; Ehab Atallah, MD, Study Chair — Medical College of Wisconsin adn Froedtert Hospital
Locations (25):
- United States (25):
  - City of Hope, Duarte, California
  - Scripps Cancer Center-Mercy, San Diego, California
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - georgia cancer Center, Augusta, Georgia
  - Pontchartrain cancer Center, Covington, Louisiana
  - RCCA MD LLC (The Center for Cancer and Blood Disorders), Bethesda, Maryland
  - Michigan Center of Medical Research, Farmington Hills, Michigan
  - Michigan State University, Breslin Cancer Center, Lansing, Michigan
  - university of minnesota medical Center, Fairview, Minneapolis, Minnesota
  - Mercy Medical Research Institute, Springfield, Missouri
  - New Mexico Cancer care Alliance, Albuquerque, New Mexico
  - University of Rochester Medical Center, Rochester, New York
  - Stony Brook University, Stony Brook, New York
  - Duke University Medical Center, Durham, North Carolina
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - Oncology Hematology Care, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cancer Centers of Southwest Oklahoma, Lawton, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute, Tulsa, Oklahoma
  - Providence Portland Medical center, Portland, Oregon
  - UT Southwestern Medical Center, Dallas, Texas
  - UVA Health System Division of Hematology & Oncology, Charlottesville, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - Universityof Wisconsin Clinical Science Center, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Stage 1 was to be conducted in 20-40 evaluable subjects to assess if the pracinostat dose regimen resulted in a discontinuation rate that met a predefined threshold, and the observed efficacy justified expansion of enrollment in Stage 1b.
  Stage 1b was conducted to achieve a planned total enrollment of 60 subjects evaluable for efficacy, inclusive of Stage 1 and Stage 1b enrollment.
Groups:
- Stage 1a and 1b Open-label Pracinostat Plus Azacitidine: open-label single arm pracinostat plus azacitidine. Pracinostat: 45 mg administered orally 3 days each week for 3 consecutive weeks, followed by 1 week of rest, in 28-day cycles.
  In later cycles (i.e., after Cycle 4), pracinostat dose reduction to 45 mg orally 3 days each week × 2 weeks (instead of 3 weeks) or dose interruption is allowed to manage toxicity such as fatigue, gastrointestinal toxicity, or myelosuppression.
  Azacitidine: 75 mg/m2 for 7 days of each 28-day cycle. Administration will occur by subcutaneous (SC) injection, or IV infusion if SC injections are not tolerated, on one of two schedules:
  * Schedule 1 - daily therapy on Days 1 through 7
  * Schedule 2 - 5-2-2 schedule in which subjects receive azacitidine for 5 consecutive days (Days 1 through 5) with rest on Days 6 and 7, and resume azacitidine dosing the first two days of the next week (Days 8 and 9) of each 28-day cycle
  Pracinostat: 45 mg capsule
  Azacitidine: SC or IV injection
Period: Overall Study
Arm/Group | Stage 1a and 1b Open-label Pracinostat Plus Azacitidine
Started | 64
Completed | 0
Not Completed | 64
Not completed — Termination of study by Sponsor | 23
Not completed — missing | 3
Not completed — Withdrawal by Subject | 8
Not completed — multiple reasons | 30

BASELINE CHARACTERISTICS:
Arm/Group | Stage 1a and 1b Open-label Pracinostat Plus Azacitidine
Number analyzed (Participants) | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (8.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 57
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 57
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 64
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] | 30.53 (5.88)

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Percentage of subjects with confirmed complete remission (CR), partial remission (PR) and marrow CR, as per modified International Working Group (IWG) criteria:
  CR: Bone marrow: ≤5% myeloblasts with normal maturation of all cell lines; Peripheral blood Hemoglobin (Hb) ≥11 g/dL; Platelets ≥100 × 10^9/L; Neutrophils ≥1.0 × 10^9/L; Blasts 0%.
  PR: All CR criteria if abnormal before treatment except: Bone marrow blasts decreased by ≥ 50% over pre-treatment but still >5%; Cellularity and morphology not relevant Marrow CR: Bone marrow: ≤5% myeloblasts and decrease by ≥50% over pre-treatment
Time Frame: 36 months
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Stage 1a and 1b Open-label Pracinostat Plus Azacitidine
Number analyzed (Participants) | 64
percentage of subjects | 35.9 [24.3 to 48.9]

2. Secondary Outcome: Complete Response (CR) Rate
Description: Percentage of subjects with confirmed CR (i.e., 2 CRs at least 28 days apart) as per modified IWG criteria:
  CR: Bone marrow: ≤5% myeloblasts with normal maturation of all cell lines; Peripheral blood Hb ≥11 g/dL; Platelets ≥100 × 109/L; Neutrophils ≥1.0 × 109/L; Blasts 0%.
Time Frame: 36 months
Measure: Number (95% Confidence Interval); unit: percentage of subjects with CR
Arm/Group | Stage 1a and 1b Open-label Pracinostat Plus Azacitidine
Number analyzed (Participants) | 64
percentage of subjects with CR | 35.9 [24.3 to 48.9]

3. Secondary Outcome: Overall Hematologic Improvement (HI) Response Rate
Description: Percentage of subjects demonstrating major hematologic improvement according to modified IWG:
  Erythroid response (pre-treatment, <11 g/dL): Hb increase by ≥1.5 g/dL; Relevant reduction of units of RBC transfusions by an absolute number of at least 4 RBC transfusions/8 weeks compared with the pre-treatment transfusion number in the previous 8 weeks. Only RBC transfusions given for a Hb of ≤9.0 g/dL pre-treatment will count in the RBC transfusion response evaluation.
  Platelet response (pre-treatment, <100 × 10^9/L): Absolute increase of ≥30 × 10^9/L for patients starting with >20 × 10^9/L platelets; Increase from <20 × 10^9/L to >20 × 10^9/L and by at least 100%.
  Neutrophil response (pre-treatment, <1.0 × 10^9/L): At least 100% increase and an absolute increase >0.5 × 10^9/L.
  Progression or relapse after HI: at least 1 of the following:
  * At least 50% decrement from maximum response levels in granulocytes or platelets
  * Reduction in Hb by≥1.5 g/dL
  * Transfusion dependence
Time Frame: 36 months
Measure: Number (95% Confidence Interval); unit: percentage of subjects with HI
Arm/Group | Stage 1a and 1b Open-label Pracinostat Plus Azacitidine
Number analyzed (Participants) | 63
percentage of subjects with HI | 71.4 [58.7 to 82.1]

4. Secondary Outcome: Clinical Benefit Rate
Description: Percentage of subjects with confirmed CR, PR, Marrow CR, and HI with clinical benefit rate, defines as rate of CR + PR + HI + Marrow CR. All subjects who achieve hematologic CR, PR, marrow CR, or hematologic improvement on the erythrocytic lineage per modified IWG response criteria will be considered responders
Time Frame: 36 months
Measure: Number (95% Confidence Interval); unit: percentage of subjects with benefit rate
Arm/Group | Stage 1a and 1b Open-label Pracinostat Plus Azacitidine
Number analyzed (Participants) | 64
percentage of subjects with benefit rate | 78.1 [66.0 to 87.5]

5. Secondary Outcome: Rate of Cytogenetic CR
Description: Percentage of subjects with confirmed CR by cytogenetic assessment. Complete cytogenetic response is defined per modified IWG response criteria:
  Complete: Disappearance of the chromosomal abnormality without appearance of new ones Partial: At least 50% reduction of the chromosomal abnormality
Time Frame: 36 months
Measure: Number (95% Confidence Interval); unit: percentage of subjects with cCR
Arm/Group | Stage 1a and 1b Open-label Pracinostat Plus Azacitidine
Number analyzed (Participants) | 64
percentage of subjects with cCR | 46.9 [34.3 to 59.8]

6. Secondary Outcome: Duration of Response (DoR)
Description: For subjects who have achieved CR, PR, Marrow CR, or HI, DoR is defined as the time from the initial determination of response to the time of disease progression or death on study, whichever occurs first.
Time Frame: 36 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stage 1a and 1b Open-label Pracinostat Plus Azacitidine
Number analyzed (Participants) | 59
months | 15.67 [9.00 to 22.11]

7. Secondary Outcome: Rate of Leukemic Transformation
Description: Percentage of subjects with leukemic transformation at landmark time point of 6 months
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Stage 1a and 1b Open-label Pracinostat Plus Azacitidine
Number analyzed (Participants) | 59
percentage of subjects | 5.4 [1.8 to 15.8]

8. Secondary Outcome: Event-free Survival (EFS)
Description: time from the first day of study drug administration (Day 1) to failure or death from any cause
Time Frame: 36 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stage 1a and 1b Open-label Pracinostat Plus Azacitidine
Number analyzed (Participants) | 59
months | 17.05 [11.50 to 21.95]

9. Secondary Outcome: Progression-free Survival (PFS)
Description: time from the first day of study drug administration (Day 1) to disease recurrence or progression as defined by the IWG criteria, or death on study:
  Disease progression for subjects with:
  Less than 5% blasts: ≥50% increase in blasts to >5% blasts 5%-10% blasts: ≥50% increase to >10% blasts 10%-20% blasts: ≥50% increase to >20% blasts 20%-30% blasts: ≥50% increase to >30% blasts
  Any of the following:
  At least 50% decrement from maximum remission/response in granulocytes or platelets Reduction in Hb by ≥2 g/dL Transfusion dependence
Time Frame: 36 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stage 1a and 1b Open-label Pracinostat Plus Azacitidine
Number analyzed (Participants) | 64
months | 16.43 [11.33 to 22.57]

10. Secondary Outcome: Overall Survival (OS)
Description: time from the first day of study drug administration (Day 1) to death on study
Time Frame: form day 1 to death on study, assessed up to 36 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stage 1a and 1b Open-label Pracinostat Plus Azacitidine
Number analyzed (Participants) | 64
months | 23.56 [16.49 to 30.26]

11. Secondary Outcome: Rate of Leukemic Transformation
Description: Percentage of subjects with leukemic transformation at landmark time point of 12 months
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Stage 1a and 1b Open-label Pracinostat Plus Azacitidine
Number analyzed (Participants) | 59
percentage of subjects | 9.5 [3.3 to 25.4]

12. Secondary Outcome: Rate of Leukemic Transformation
Description: Percentage of subjects with leukemic transformation at landmark time point of 18 months
Time Frame: 18 months
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Stage 1a and 1b Open-label Pracinostat Plus Azacitidine
Number analyzed (Participants) | 59
percentage of subjects | 13.8 [5.5 to 32.4]

13. Secondary Outcome: Rate of Leukemic Transformation
Description: Percentage of subjects with leukemic transformation at landmark time point of 24 months
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Stage 1a and 1b Open-label Pracinostat Plus Azacitidine
Number analyzed (Participants) | 59
percentage of subjects | 21.6 [8.8 to 47.3]

ADVERSE EVENTS:
Time Frame: All AEs regardless of seriousness or relationship to pracinostat or azacitidine, from the start of study drug treatment until 30 calendar days after discontinuation or completion of treatment as defined by the clinical study for that subject, have been recorded.
Arm/Group | Stage 1a and 1b Open-label Pracinostat Plus Azacitidine
All-Cause Mortality (participants affected / at risk) | 5/64
Serious Adverse Events (participants affected / at risk) | 45/64
Other Adverse Events (participants affected / at risk) | 64/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1a and 1b Open-label Pracinostat Plus Azacitidine (N=64)
Febrile neutropenia (Blood and lymphatic system disorders) | 17
Pancytopenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Acute coronary syndrome (Cardiac disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 2
Sinus tachycardia (Cardiac disorders) | 1
Anal fissure (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Proctitis (Gastrointestinal disorders) | 1
Rectal ulcer (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 2
Malaise (General disorders) | 1
Pyrexia (General disorders) | 1
Abscess limb (Infections and infestations) | 1
Anal abscess (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Clostridial sepsis (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Escherichia sepsis (Infections and infestations) | 1
Fungal oesophagitis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Lung infection (Infections and infestations) | 3
Perirectal abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 6
Pseudomonal sepsis (Infections and infestations) | 1
Respiratory tract infection viral (Infections and infestations) | 1
Sepsis (Infections and infestations) | 5
Sialoadenitis (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Streptococcal sepsis (Infections and infestations) | 1
Vascular access site infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Electrocardiogram qt prolonged (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperinsulinaemic hypoglycaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Presyncope (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 1
Mania (Psychiatric disorders) | 1
Mental disorder (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1a and 1b Open-label Pracinostat Plus Azacitidine (N=64)
Anaemia (Blood and lymphatic system disorders) | 31
Febrile neutropenia (Blood and lymphatic system disorders) | 23
Leukopenia (Blood and lymphatic system disorders) | 7
Neutropenia (Blood and lymphatic system disorders) | 9
Pancytopenia (Blood and lymphatic system disorders) | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 18
Tachycardia (Cardiac disorders) | 7
Ear pain (Ear and labyrinth disorders) | 4
Dry eye (Eye disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 33
Diarrhoea (Gastrointestinal disorders) | 21
Dry mouth (Gastrointestinal disorders) | 7
Dyspepsia (Gastrointestinal disorders) | 6
Dysphagia (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 34
Oral pain (Gastrointestinal disorders) | 5
Proctalgia (Gastrointestinal disorders) | 4
Tongue discolouration (Gastrointestinal disorders) | 14
Vomiting (Gastrointestinal disorders) | 16
Asthenia (General disorders) | 6
Chest pain (General disorders) | 5
Chills (General disorders) | 9
Fatigue (General disorders) | 29
Injection site reaction (General disorders) | 7
Oedema peripheral (General disorders) | 23
Pyrexia (General disorders) | 12
Lung infection (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 8
Sepsis (Infections and infestations) | 6
Sinusitis (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 4
Contusion (Injury, poisoning and procedural complications) | 10
Fall (Injury, poisoning and procedural complications) | 10
Blood alkaline phosphatase increased (Investigations) | 4
Blood creatinine increased (Investigations) | 8
International normalised ratio increased (Investigations) | 5
Lymphocyte count decreased (Investigations) | 5
Neutrophil count decreased (Investigations) | 34
Weight decreased (Investigations) | 7
White blood cell count decreased (Investigations) | 14
Decreased appetite (Metabolism and nutrition disorders) | 26
Dehydration (Metabolism and nutrition disorders) | 10
Hyperglycaemia (Metabolism and nutrition disorders) | 8
Hypoalbuminaemia (Metabolism and nutrition disorders) | 18
Hypocalcaemia (Metabolism and nutrition disorders) | 9
Hypoglycaemia (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 16
Hyponatraemia (Metabolism and nutrition disorders) | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 13
Arthritis (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 8
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9
Dizziness (Nervous system disorders) | 19
Dysgeusia (Nervous system disorders) | 7
Headache (Nervous system disorders) | 8
Presyncope (Nervous system disorders) | 4
Syncope (Nervous system disorders) | 4
Tremor (Nervous system disorders) | 7
Anxiety (Psychiatric disorders) | 10
Confusional state (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 12
Acute kidney injury (Renal and urinary disorders) | 9
Pollakiuria (Renal and urinary disorders) | 4
Urinary retention (Renal and urinary disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 15
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 10
Papule (Skin and subcutaneous tissue disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 11
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10
Hypertension (Vascular disorders) | 8
Hypotension (Vascular disorders) | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-06-25): https://cdn.clinicaltrials.gov/large-docs/04/NCT03151304/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-28): https://cdn.clinicaltrials.gov/large-docs/04/NCT03151304/SAP_001.pdf